CLINICAL TRIAL: NCT02642458
Title: Pertuzumab in First Line Treatment of HER2-positive Metastatic Breast Cancer Patients: A Cohort Study of Patients Treated Either With Docetaxel and Trastuzumab or Docetaxel, Trastuzumab and Pertuzumab
Brief Title: Pertuzumab in First Line Treatment of HER2-positive Metastatic Breast Cancer Patients
Acronym: PerFECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: SEN2015-02
Record Dates: First submitted 2015-12-09; First posted 2015-12-30 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- trastuzumab plus chemotherapy: Treatment with trastuzumab plus chemotherapie as first line therapy, administered intravenously/subcutaneously in a three weekly frequency. Docetaxel is recommended as chemotherapy, however, any treatment choice or change in regimen is performed at the discretion of the treating physician.
- pertuzumab plus trastuzumab plus chemotherapy: Treatment with with pertuzumab plus trastuzumab plus chemotherapy as first line therapy, administered intravenously/subcutaneously in a three weekly frequency. Docetaxel is recommended as chemotherapy, however, any treatment choice or change in regimen is performed at the discretion of the treating physician.

SUMMARY:
Despite the clear benefit of a combination therapy of pertuzumab plus trastuzumab plus docetaxel when compared with a combination therapy of trastuzumab and docetaxel the study populations of the CLEOPATRA trial might be slightly different from a patient population, in which pertuzumab, plus trastuzumab plus chemotherapy or trastuzumab plus chemotherapy are applied in routine clinical practice.

This non-interventional approach aims to confirm the clinically relevant outcomes shown in the phase III CLEOPATRA study in patients with advanced HER2-positive breast cancer in routine practice. Docetaxel is recommended as chemotherapy, however, any treatment choice or change in regimen is performed at the discretion of the treating physician.

Data on efficacy, safety, tolerability and quality of life will be documented for this purpose. Following the recommendations as laid down in guidelines for treatment of breast cancer, the quality of life of patients will be assessed on a regular basis.

DETAILED DESCRIPTION:
Breast cancer is the commonest cancer in women worldwide with an estimated 1.4 million new diagnoses in 2008 and 1.6 million cases estimated for 2015. In 2008 breast cancer was responsible for approximately 23% of all new cancer diagnoses in women. It is also the commonest cause of cancer deaths in women worldwide: in 2008 some 458,500 women died from breast cancer, with a further 538,500 projected for 2015.

In developed countries most breast cancers (in 94%-95% of patients in the EU and USA) are diagnosed while the tumour is confined to the breast - with or without locoregional lymph node involvement. At this early breast cancer (EBC) stage the disease is normally operable and can be treated curatively. Metastatic breast cancer (MBC) is less common and occurs in 5%-6% of newly diagnosed cases. Despite advances in the treatment of EBC approximately 30% of women develop local recurrence or metastases. In the USA and Europe patients with MBC survive for a mean 24 months and have a 5 year survival rate of 18%-23%.

Between 18% and 20% of breast cancers show HER2 amplification and/or HER2 receptor overexpression. Such patients have a poor prognosis on conventional treatment. The HER2 receptor is a protein belonging to the epidermal growth factor receptor (EGFR) family. The HER family consists of four structurally similar receptors - HER1/EGFR, HER2, HER3, HER4 - and regulates cell processes such as differentiation, invasion, proliferation, neoangiogenesis, survival and metastatic potential. In breast cancer HER2 positivity is associated with more aggressive tumours, higher relapse rates, lower and shorter treatment response and increased mortality.

Systemic treatment options in MBC include chemotherapy along with hormonal and targeted approaches. Tumor properties and patient-specific factors determine the choice of treatment.

In HER2-positive MBC trastuzumab for many years was the reference first-line treatment. Treatment-naive HER2-positive patients with MBC treated with trastuzumab and taxane chemotherapy showed significantly longer median time to progression (TTP), higher objective response rates (ORR) and longer median response and median survival than patients treated with chemotherapy alone. Although trastuzumab has proved effective in combination with chemotherapy in the first-line treatment of patients with HER2-positive MBC, approximately 50% of patients experience disease progression within one year of starting treatment. Mean survival in HER2-positive patients in the pivotal studies of trastuzumab in combination with a taxane was 24.8 and 31.2 months.

Therefore there is high medical need for novel HER2-targeted therapies to improve survival outcomes in patients with HER2-positive MBC.

An essential step in activating downstream signalling pathways is homo or heterodimerisation of the HER2 receptor with the other member of the HER family. Inhibition of HER2 dimerisation inhibits the downstream signalling pathways that mediate cancer cell proliferation and survival. Pertuzumab, a humanised monoclonal antibody, is the first HER2 dimerisation inhibitor (HDI). It binds specifically to the extracellular dimerisation domain of the HER2 receptor, thereby inhibiting ligand-dependent heterodimerisation of the receptor with other HER family members. Pertuzumab actually inhibits ligand-activated intracellular signal transduction in two main signalling pathways - the mitogen-activated protein kinase (MAPK) pathway and the phosphoinositide-3-kinase (PI3K) pathway. Inhibition of these signalling pathways can arrest cell growth and cause apoptosis. Pertuzumab also mediates antibody-dependent cell-mediated cytotoxicity (ADCC). Pertuzumab and trastuzumab bind to different epitopes on the HER2 receptor. Their mechanisms of action complement each other to ensure more comprehensive blockade of HER2-dependent signalling pathways.

The phase III, multicentre, randomised, double-blind and placebo-controlled clinical CLEOPATRA trial compared pertuzumab plus trastuzumab plus docetaxel vs placebo plus trastuzumab plus docetaxel in 808 patients with HER2-positive metastatic, locally recurrentor inoperable breast cancer. Patients may have received one hormonal treatment for metastatic breast cancer before randomization. Patients may have received adjuvant or neoadjuvant chemotherapy with or without trastuzumab before randomization, with an interval of at least 12 months between completion of the adjuvant or neoadjuvant therapy and the diagnosis of metastatic breast cancer. Randomised patients were stratified by previous treatment status (with or without previous adjuvant/neoadjuvant therapy) and geographic location (Europe, North America, South America and Asia). Pertuzumab was given intravenously at a starting dose of 840 mg followed by a dose of 420 mg every 3 weeks. Trastuzumab was given intravenously at a starting dose of 8 mg/kg followed by a dose of 6 mg/kg every 3 weeks. Patients were treated with pertuzumab plus trastuzumab until disease progression, withdrawal of consent to participation or the development of uncontrollable toxicity. Docetaxel was given as an intravenous infusion at a starting dose of 75 mg/m² every 3 weeks for at least 6 cycles. If the starting dose was well-tolerated, the dose of docetaxel could be increased up to 100 mg/m² at the investigator's discretion.

The primary study endpoint was progression-free survival (PFS), assessed by an independent review facility (IRF) and defined as the interval between randomisation and disease progression or death (from any cause), where death occurred within 18 weeks of the last disease assessment. The secondary endpoints were overall survival (OS), (investigator-rated) PFS, objective response rate (ORR), duration of response and time to progression (TTP).

Demographic characteristics were evenly balanced (mean age was 54 years, most [59%] were Caucasian and all but two were female). In each treatment group approximately half the patients had hormone (estrogen or progesterone) receptor-positive disease and had received previous adjuvant or neoadjuvant therapy (184 patients [45.8%] in the pertuzumab group vs 192 patients [47.3%] in the placebo group). Most (37.3% and 40.4%, respectively) had previously received anthracyclines and approximately 10% had previously received trastuzumab (11.7% and 10.1%). A total 43% of patients from both groups had received prior radiotherapy. The mean baseline left ventricular ejection fraction (LVEF) was 64.8% in the pertuzumab group and 65.6% in the placebo group (median 65.0%, range 50%-88% in the two groups).

The CLEOPATRA study showed statistically significant improvement of IRF-rated PFS in the pertuzumab group vs placebo (hazard ratio [HR]=0.62; 95% CI=0.51; 0.75, p<0.0001) and an increase in median PFS of 6.1 months. Median PFS was 18.5 months in the pertuzumab group vs 12.4 months in the placebo group. Moreover, CLEOPATRA showed statistically significant improvement of overall survival in the pertuzumab group vs placebo (hazard ratio [HR]=0.68; 95% CI=0.56; 0.84, p<0.0002) and an increase in median OS of 15.7 months. Median OS was 56.5 months in the pertuzumab group vs 40.8 months in the placebo group.

Despite the clear benefit of a combination therapy of pertuzumab plus trastuzumab plus docetaxel when compared with a combination therapy of trastuzumab and docetaxel the study populations of the CLEOPATRA study might be slightly different from a patient population, in which pertuzumab, plus trastuzumab plus docetaxel or trastuzumab plus docetaxel are applied in routine clinical practice.

This non-interventional approach aims to confirm the clinically relevant outcomes shown in the phase III CLEOPATRA study in patients with advanced HER2-positive breast cancer in routine practice. Data on efficacy, safety, tolerability and quality of life will be documented for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Adult breast cancer patients (age ≥18 years)
* Patients with metastatic or locally advanced, unresectable HER2-positive breast cancer proven by clinical measures (i.e. standard imaging) in first line treatment (Locally recurrent disease must not be amenable to resection with curative intent)
* Patients who are eligible for treatment with trastuzumab plus chemotherapy or pertuzumab plus trastuzumab plus chemotherapy as first line therapy, administered intravenously in a three weekly frequency, according to each center's medical practice. The first line anti-HER2 treatment must not have started more than 28 days before study entry.
* No prior chemotherapy or HER2-directed therapy for metastatic or locally advanced disease, prior therapy for early breast cancer (eBC) is allowed
* Signed informed consent prior to onset of documentation.

Exclusion Criteria:

• Patients who are not eligible for observation due to severe comorbidities or unavailability according to the treating physician

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted as an open registry, therefore there will be no restriction in the number of patients to be included.
  The assignment of the patient to a particular treatment falls within current practice and the prescription of the medicine is clearly separated from the decision to include the patient in the non-interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
progression free survival rate | At 12 months or month 36
  The primary objective of this study is to assess the progression free survival rate at month 12 for both treatment cohorts in routine clinical practice treated with either pertuzumab plus trastuzumab plus docetaxel or trastuzumab plus docetaxel.

SECONDARY OUTCOMES:
Progression free survival | Timepoint of progression or month 36
  Progression free survival (PFS) is defined as the time interval from start of therapy until progression proven with clinical measures according to expertise and daily clinical routine or death from any cause, whichever comes first.
Overall response rate | Timepoint of progression or month 36
  Overall response rate (ORR): Rate of complete (CR) and partial responses (PR) in patients. Response to treatment (CR, PR, SD, and PD) will be assessed by the treating physician and evaluated according to expertise and daily clinical routine. Underlying method of response assessment will be captured.
Quality of life (EORTC QLQ-C30) | At 12 months
  Quality of life (QoL) will be assessed by the EORTC QLQ-C30 (Version 3.0) within the first 12 months of first line treatment either with docetaxel and trastuzumab or docetaxel, trastuzumab and pertuzumab. The minimum target return rate for PRO questionnaires is 70% defined as at least 70% of patients having completed the PRO questionnaires at all collection time points.
Incidence of adverse events and serious adverse events will be documented | up 36 month
  Incidence of adverse events and serious adverse events will be reported according to NCI Common Toxicity Criteria Version 4.03.
Quality of life (EORTC QLQ-BR23) | At 12 months
  Quality of life (QoL) will be assessed by the EORTC QLQ-BR23 (Version 1.0) within the first 12 months of first line treatment either with docetaxel and trastuzumab or docetaxel, trastuzumab and pertuzumab. The minimum target return rate for PRO questionnaires is 70% defined as at least 70% of patients having completed the PRO questionnaires at all collection time points.

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Wallwiener, Prof. Dr., Study Director — Universitätsfrauenklinik Tübingen; Peter Fasching, Prof. Dr., Principal Investigator — Frauenklinik des Universitätsklinikums Erlangen; Sara Brucker, Prof. Dr., Study Director — Universitätsklinikum Tübingen Universitäts-Frauenklinik
Locations (37):
- Germany (37):
  - Klinikum für Frauenheilkunde und Geburtshilfe Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Onkologische Schwerpunktpraxis Heidelberg, Heidelberg, Baden-Wurttemberg
  - NCT Heidelberg, Heidelberg, Baden-Wurttemberg
  - Frauenklinik des Städtischen Klinikums, Karlsruhe, Baden-Wurttemberg
  - St. Vicentius Kliniken Karlsruhe gAG Frauenklininik, Karlsruhe, Baden-Wurttemberg
  - Ortenau Klinikum Lahr-Ettenheim, Lahr, Baden-Wurttemberg
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Klinikum Mannheim, Universitäts-Frauenklinik, Mannheim, Baden-Wurttemberg
  - Universitätsfrauenklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Onkokom GbR, Altötting, Bavaria
  - MVZ Amberg, Amberg, Bavaria
  - Klinikum Augsburg Frauenklinik, Augsburg, Bavaria
  - Rottal-Inn-Kliniken GmbH, Eggenfelden, Bavaria
  - Universitätsfrauenklinik Erlangen, Erlangen, Bavaria
  - Hämatologisch-Onkologische Praxis, Kronach, Bavaria
  - Klinikum Nürnberg AöR, Nuremberg, Bavaria
  - Hochschulklinikum der Med. Hochschule Brandenburg, Neuruppin, Brandenburg
  - g.SUND Gynäkologie Kompetenzzentrum, Stralsund, Brandenburg
  - Klinikum Darmstadt, Frauenklinik, Darmstadt, Hesse
  - Zentrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main, Hesse
  - MVZ Onkologische Kooperation Harz Onkologische Schwerpunktpraxis, Goslar, Hesse
  - Frauenklinik Wetzlar, Wetzlar, Hesse
  - Agaplesion Diakonieklinikum Rotenburg/Wümme gGmbH, Rotenburg (Wümme), Lower Saxony
  - Gemeinschaftspraxis f. Hämatologie u. Onkologie, Westerstede, Lower Saxony
  - Facharztzentrum am Schloß, Wolfenbüttel, Lower Saxony
  - MarienHospital Onkologische Praxis, Bonn, North Rhine-Westphalia
  - Marienhospital Bottrop gGmbH, Bottrop, North Rhine-Westphalia
  - Institut für Versorgungsforschung in der Onkologie, Cologne, North Rhine-Westphalia
  - Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe des Universitätsklinikums Köln Brustzentrum, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Schwerpunktpraxis für Hämatologie und Onkologie Hansen/Reeb/Pfitzner-Dempfle/Stehle, Kaiserslautern, Rhineland-Palatinate
  - Klinikum Chemnitz gGmbH Frauenklinik, Chemnitz, Saxony
  - Onkologische Gemeinschaftspraxis Dresden, Dresden, Saxony
  - Universitäres Krebszentrum Leipzig, Leipzig, Saxony
  - Gemeinschaftspraxis, Halle, Saxony-Anhalt
  - MediOnko-Institut GbT, Berlin
  - Onkologisch-Hämatologische Schwerpunktpraxis, Bremen

IPD SHARING:
Plan to Share IPD: Undecided